CLINICAL TRIAL: NCT01089361
Title: Immunomodulatory Properties of Ketamine in Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Talmor, Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P000259
Record Dates: First submitted 2010-03-12; First posted 2010-03-18 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Sepsis
Keywords: systemic inflammatory syndrome; sepsis syndrome; septic shock; Cytokine; Ketamine
MeSH Terms: conditions — Sepsis; Systemic Inflammatory Response Syndrome; Shock, Septic | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline placebo (Placebo Comparator): The control group will receive 0.25mg/kg of normal saline over a period of one hour followed by a continuous infusion of normal saline at 0.1 mg/kg/hr for a further 23 hours.
  Interventions: Drug: Normal Saline placebo
- Ketamine (Experimental): The treatment group will receive 0.25mg/kg of ketamine over a period of one hour followed by a continuous infusion of ketamine at 0.1 mg/kg/hr for a further 23 hours.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — The treatment group will receive 0.25mg/kg of ketamine over a period of one hour followed by a continuous infusion of ketamine at 0.1 mg/kg/hr for a further 23 hours.
  Other Names: Ketamine Hydrochloride; Ketalar
  Arms: Ketamine
Drug: Normal Saline placebo — The control group will receive 0.25mg/kg of normal saline over a period of one hour followed by a continuous infusion of normal saline at 0.1 mg/kg/hr for a further 23 hours.
  Other Names: 0.9% Sodium Chloride Solution
  Arms: Normal saline placebo

SUMMARY:
The aim of the study is to assess the effect of short-term infusion of ketamine at analgesic dosage on the immune response, morbidity and mortality among patients suffering from septic shock. We hypothesize that ketamine will modulate the cytokine response to sepsis and reduce morbidity and mortality.

DETAILED DESCRIPTION:
1. Basic design A randomized placebo controlled trial of low dose ketamine in patients with severe sepsis in the ICU.
2. Assembly of Subjects Patients meeting the ACCP/ SCCM definition of severe sepsis will be enrolled in the study5. These patients should have a known or suspected source of infection based on the clinical data at the time of screening. They must exhibit 3 or more of the following signs of clinical inflammation

   * Core temperature < 36ºC or > 38ºC.
   * Heart rate of 90 or greater not explained by another medical condition.
   * A respiratory rate of > 20 min-1, a PaCO2 < 32min-1 or the need for mechanical ventilation.
   * A white cell count of < 4000 cell/ml or > 12000 cells/ml or a WBC showing greater then 10% immature neutrophils.

   In addition the patient will have to be within 12 hours of the development of one or more organ dysfunctions as outlined in Bone et al 5.

   Several exclusion criteria will be in place to safeguard patient's safety 11. Patients with closed head trauma or with increased intracranial pressure will be excluded. Patients with a history of psychotic mental disease will also be excluded as they may be at risk for relapse following administration of ketamine.
3. Exposures Patients will be randomized into a treatment group and a control group. The treatment group will receive 0.25mg/kg of ketamine over a period of one hour followed by a continuous infusion of ketamine at 0.1 mg/kg/hr for a further 23 hours. To help insure protocol compliance and safeguard patient care, a member of the study team will be present at the time the study drug infusion is started, and will also contact the clinical team when the infusion is due to be terminated. The dose of the ketamine is considered analgesic not anesthetic in nature and follows general practice in pain management 11. The control group will receive a similar volume of normal saline as a placebo. Additionally all patients enrolled in the study will receive lorazepam 1mg every 6 hours to further lower the risk of side effect from ketamine. Patients, staff and investigators will all be blinded to the treatment groups. All other care, including the need for further sedation, will be according to unit protocols.

   Prior to administration of the study drug a 10cc sample of the patient's blood will be drawn and frozen for later analysis. 2 hours after starting infusion another 10ml of blood will be obtained. Following 24 hour infusion of ketamine, blood samples will be drawn each day, for the following 7 days, processed and frozen.

   Patient demographic and clinical data will be collected on admission to the study and daily follow-up. Particular attention will be paid to calculation of the patient's APACHE II/MODS score on the day of admission and on the following days22. This will allow us to compare severity of disease in a potentially heterogeneous ICU patient population. We will also monitor use of the vasopressors, additional pain and sedative medication and physiological parameters (BP, HR, Sat, ABG, LFT, lactic acid) in studied population before and after administration of the drug. The adverse effect of ketamine will assessed by using delirium questionnaire and special chart designed to capture the emergence of side effect (delirium, psychosis, others).
4. Outcomes and their measurement The primary outcome of the study will be serum levels of IL-6, IL-10 and TNFα and other cytokines over the first 7 days of admission. Measurement of cytokine levels will be done using enzyme linked immunoassay, or with flow cytometry at the end of the study by at researcher who will be blinded to the study groups. We also plan to separate leukocytes for further studies of mRNA levels to corroborate serum cytokine levels with activity of mRNA.

   Secondary outcomes will include adverse effects attributable to ketamine, organ failures, daily APACHE scores, length of ICU stay and 28 day mortality. A clinical research associate will carry out a daily patient assessment. This investigator will be blinded to the treatment groups. Data will be collected on a patient study chart. In addition to the incidence of organ dysfunction, death and length of stay, specific information will be gathered to assess patient's level of conscience, possible dreams or hallucinations and other effects, which may be attributable to ketamine.
5. Substudy of serum samples We plan to perform real-time quantitative PCR analyses on the existing serum samples for the presence of bacterial and mitochondrial DNA on the samples. We will use primers targeting bacterial 16S-rRNA consensus areas and primers targeting gram-positive (S. Aureus), gram-negative (e. coli) and anaerobic (B. Fragilis) species. These tests may be able to accurately discriminate between systemic inflammation ("SIRS") due to invasive bacterial infections from SIRS due to tissue injury than do conventional bacteriologic analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the ACCP/ SCCM definition of severe sepsis will be enrolled in the study. These patients should have a known or suspected source of infection.
* Patients within 12 hours of the development of one or more organ dysfunctions
* Patients must exhibit 3 or more of the following signs of clinical inflammation:

  * Core temperature < 36ºC or > 38ºC.
  * Heart rate of 90 or greater not explained by another medical condition.
  * A respiratory rate of > 20 min-1, a PaCO2 < 32min-1 or the need for mechanical ventilation.
  * A white blood cell count of < 4000 cell/ml or > 12000 cells/ml or a WBC showing greater then 10% immature neutrophils.

Exclusion Criteria:

* pregnant
* increased intracranial pressure or closed head injury
* history of psychotic mental disease
* receiving Continuous Veno - Venous Hemofiltration

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calandra T, Bochud PY, Heumann D. Cytokines in septic shock. Curr Clin Top Infect Dis. 2002;22:1-23. No abstract available. PMID 12520644
- [Background] Laudanski K, Miller-Graziano C, Xiao W, Mindrinos MN, Richards DR, De A, Moldawer LL, Maier RV, Bankey P, Baker HV, Brownstein BH, Cobb JP, Calvano SE, Davis RW, Tompkins RG. Cell-specific expression and pathway analyses reveal alterations in trauma-related human T cell and monocyte pathways. Proc Natl Acad Sci U S A. 2006 Oct 17;103(42):15564-9. doi: 10.1073/pnas.0607028103. Epub 2006 Oct 10. PMID 17032758
- [Background] Kawasaki T, Ogata M, Kawasaki C, Ogata J, Inoue Y, Shigematsu A. Ketamine suppresses proinflammatory cytokine production in human whole blood in vitro. Anesth Analg. 1999 Sep;89(3):665-9. doi: 10.1097/00000539-199909000-00024. PMID 10475301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 2009 and 2010 from the ICU.
Pre-assignment Details: All patients who consented were randomized to treatment or placebo.
Groups:
- Normal Saline: The control group will receive 0.25mg/kg of normal saline over a period of one hour followed by a continuous infusion of normal saline at 0.1 mg/kg/hr for a further 23 hours.
Period: Overall Study
Arm/Group | Normal Saline | Ketamine
Started | 9 | 10
Completed | 8 | 10
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Ketamine | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (19) | 60 (11) | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of IL-6, IL-10 and TNFα
Time Frame: first 7 days of admission, Baseline and Day 7 reported
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 8 | 10
pg/mL
  Baseline IL-10 | 28 [8.1 to 246.9] | 16 [12.2 to 19.6]
  Day 7 IL-10 | 9.3 [4.7 to 12.9] | 6.3 [5 to 10.5]
  Baseline IL-6 | 3227.7 [512 to 7205.7] | 613.8 [320.8 to 3190.5]
  Day 7 IL-6 | 322.8 [96.8 to 428] | 266.2 [56.3 to 285.8]
  Baseline TNF-alpha | 2.5 [1.5 to 6.2] | 7.1 [3.2 to 7.9]
  Day 7 TNF-alpha | 2 [1.2 to 3.1] | 6.3 [2.4 to 15.4]

2. Secondary Outcome: Adverse Effects Attributable to Ketamine
Time Frame: 7 days
Measure: Number; unit: adverse events
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 9 | 10
adverse events | 0 | 2

3. Secondary Outcome: Organ Failures
Description: Incidence of new organ failure as detected by Sequential Organ Failure Assessment [SOFA] score. Definitions are as follows. Central nervous system: delirium, coma, uncontrollable seizures, ICP>20cm H2O Cardiac: MAP <60mmHg, blood pressure supported with pressors, 50 > HR > 120 Respiratory: vented, RR>30, PaO2<60, PaCO2 > 55, Sat<92% Kidney: RIFLE criteria Anemia: Hct<27, transfusion of PRBC Thrombocytopenia: platelet < 50k, platelet transfusion Liver: biopsy, ALT>200, AST>200, t.bil>2.0, ALP>300 Coagulation failure: INR>2 if no anticoagulation therapy
Time Frame: 7 days
Measure: Number; unit: participants with increase in SOFA score
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 9 | 10
participants with increase in SOFA score | 3 | 2

4. Secondary Outcome: Acute Physiology and Chronic Health Evaluation (APACHE) Scores
Description: Difference in average APACHE-II score between the intervention and placebo groups. APACHE II (Acute Physiology and Chronic Health Evaluation II) is a severity of disease classification system for patients admitted to the Intensive Care Unit. It uses an integer score from 0 to 71 that is computed based on age, 12 routine physiological measurements (i.e. heart rate, temperature, laboratory values), and previous health status obtained during the first 24 hours after ICU admission. Higher scores correspond to more severe disease and a higher risk of death.
Time Frame: First 24 hours after ICU admission
Measure: Mean (Standard Deviation); unit: APACHE score
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 9 | 10
APACHE score | 25 (8) | 23 (10)

5. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 8 | 10
days | 19 (9) | 20 (9)

6. Secondary Outcome: 28 Day Mortality
Time Frame: 28 days
Measure: Number; unit: deaths
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 9 | 10
deaths | 4 | 2

7. Other Pre Specified Outcome: PCR Substudy
Description: PCR analysis on serum samples for presence of bacterial and mitochondrial DNA; This substudy was not done.
Time Frame: Daily up to 7 days
Population: Not done
Arm/Group | Normal Saline Placebo | Ketamine
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Time Frame: Seven days from enrollment.
Arm/Group | Normal Saline | Ketamine
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/10
Other Adverse Events (participants affected / at risk) | 0/9 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=9) | Ketamine (N=10)
Death (General disorders) | 4 (4) | 2 (2) — All deaths in this trial were expected based on patients' clinical course and followed withdrawal of clinical care. None were suspected of being related to trial participation.
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) — Pericardial effusion, possible tamponade. Treated with drainage.
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — Treated with antiarrythmics
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=9) | Ketamine (N=10)
Tachycardia (atrial fibrillation) (Cardiac disorders) | 0 (0) | 3 (3) — Clinically expected based on septic presentation. Treated with cardioversion and medication.
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
Salivation, excessive (Gastrointestinal disorders) | 0 (0) | 1 (1) — Possibly related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes